CLINICAL TRIAL: NCT00298870
Title: Randomized Trial for Pharmacogenomics-based Tuberculosis Therapy (RT-PGTT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG-MRT-TB-01
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2011-05

CONDITIONS: Pulmonary Tuberculosis
Keywords: pulmonary tuberculosis; isoniazid; arylamine N-acetyltransferase 2; pharmacogenomics; genetic polymorphisms; individualized medicine; drug-induced hepatotoxity
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PGx-treatment (Experimental): NAT2 genotype-guided treatment with stratified isoniazid dose (approx. 7.5 mg/kg b.w., patients homozygous for NAT2*4: rapid acetylators; 5 mg/kg, patients heterozygous for NAT2*4: intermediate acetylators; 2.5 mg/kg, patientes without NAT2*4: slow acetylators)
  Interventions: Drug: Isoniazid
- STD-treatment (Active Comparator): Treatment with conventional standard isoniazid dose (approx. 5 mg/kg b.w.)
  Interventions: Drug: isoniazed

INTERVENTIONS:
Drug: Isoniazid — Modified daily isoniazid dose : approx. 7.5 mg/kg, 5 mg/kg and 2.5 mg/kg for rapid, intermediate and slow acetylators, respectively
  Arms: PGx-treatment
Drug: isoniazed — Conventional standard daily isoniazid dose : approx. 5 mg/kg b.w. for all
  Arms: STD-treatment

SUMMARY:
The purpose of this study is to elucidate whether the individualized medicine based on NAT2 gene polymorphism could improve the safety, efficacy and economical benefits of multi-drug therapy for the pulmonary tuberculosis with isoniazid.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pulmonary tuberculosis patients
* Informed consent including pharmacogenomic analysis

Exclusion Criteria:

* Abnormal liver and kidney function test before treatment
* Long-term use of steroids and/or immunodepressants
* Inadequate clinical conditions

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2005-06

PRIMARY OUTCOMES:
The incidences of unfavorable events in two different treatment regimens based on the NAT2 gene polymorphism
  1) the incidences of drug-induced liver injury associated with INH that occurred within 8 weeks of the treatments, and 2) the incidence of early treatment failure as indicated by a persistent positive culture or no improvement in chest radiographs at the 8th week

SECONDARY OUTCOMES:
Other adversed events during the 8 weeks of the intensive phase of the anti-tuberculosis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Azuma, MD, Study Chair — Graduate School of Pharmaceutical Sciences, Osaka University
Locations (4):
- Japan (4):
  - Osaka Prefectural Medical Center for Respiratory and Allergic Diseases, Habikino, Osaka
  - Osaka Hospital, Anti-Tuberculosis Association, Osaka Branch, Neyagawa, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai, Osaka
  - National Hospital Organization Toneyama, Toyonaka, Osaka

REFERENCES:
- [Derived] Azuma J, Ohno M, Kubota R, Yokota S, Nagai T, Tsuyuguchi K, Okuda Y, Takashima T, Kamimura S, Fujio Y, Kawase I; Pharmacogenetics-based tuberculosis therapy research group. NAT2 genotype guided regimen reduces isoniazid-induced liver injury and early treatment failure in the 6-month four-drug standard treatment of tuberculosis: a randomized controlled trial for pharmacogenetics-based therapy. Eur J Clin Pharmacol. 2013 May;69(5):1091-101. doi: 10.1007/s00228-012-1429-9. Epub 2012 Nov 14. PMID 23150149